CLINICAL TRIAL: NCT02707029
Title: Clinical and Scientific Assessment of Pain and Painful Disorders
Status: Recruiting | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160077; 16-AT-0077
Record Dates: First submitted 2016-03-08; First posted 2016-03-14 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2026-01-15

CONDITIONS: Normal Physiology; Pain
Keywords: Screening Protocol; Pain; Phenotypes
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons, with or without pain disorders: Adults and adolescents with or without pain disorders.

SUMMARY:
Background:

Researchers want to better understand pain by studying people with and without different kinds of pain. To do this, researchers will expose people to pleasant and unpleasant sensations. They will ask them questions about their pain. Researchers also want to see if these people are eligible for other research studies at the National Center for Complementary and Integrative Health.

Objectives:

To study the experience of pain. Also to find people eligible to join other NIH studies.

Eligibility:

People 12 years and older with and without pain disorders.

Design:

Participants will be screened by phone.

Participants will have one required visit lasting about 2 hours. This may include:

* Medical history
* Physical exam
* Questionnaires about themselves and their pain experience
* Blood and urine tests
* MRI: They will lie on a table that slides into a cylinder. They will feel different sensations while completing tasks on a computer. This lasts 15 minutes to 2 hours.
* Quantitative sensory testing: They will be exposed to different pictures, sounds, tastes, and smells. They will also be exposed to pleasant and unpleasant sensations. These could include:

  * Burning, itching, or cold sensations
  * Pinpricks
  * Pressure and pinches
* Electrocardiogram: Stickers on the chest record heart activity.
* Straps placed around the chest to measure breathing.
* Small sensors on the fingers or palms to measure pulse and sweating.

Participants may have up to 12 other outpatient study visits.

Participants may be recorded at the visits.

DETAILED DESCRIPTION:
Objective:

The purpose of this study is to allow for the deep, broad, and targeted phenotyping of persons with or without pain disorders. This protocol will enable NCCIH investigators to describe the clinical aspects of pain disorders, collect scientific measurements for the purpose of making deep phenotypic descriptions, and use the collected data to perform descriptive analyses of pain disorders. The study will also facilitate obtaining information relevant to determining if a person is potentially eligible to participate in other research protocols at NIH, in particular those of the Laboratory of Clinical Investigation (LCI) at the National Center for Complementary and Integrative Health (NCCIH). The specific goals of this protocol are the following:

Research:

* To enable the clinical description and phenotyping of research participants, in particular those with pain disorders.
* To facilitate obtaining information relevant to determining potential eligibility of consenting participants to participate in other IRB-approved NIH protocols that focus on pain and related disorders.
* To perform descriptive analyses of painful experiences within discrete pain disorders.

Study Population: The study population will consist of up to 10,000 persons with or without pain disorders, who seek to participate in research protocols at NIH, primarily those sponsored by NCCIH Division of Intramural Research investigators. Human beings of adolescence age or older (>= 12 years) that are willing to provide assent and/or consent may participate in the study. This protocol is open to participants of any ethnicity, gender, or nationality.

Design:

The protocol is designed as a cross-sectional observational study. Participants will initially undergo an informed consent process and a core phenotyping evaluation, which includes a clinical evaluation from a Licensed Independent Practitioner (LIP) and questionnaires. Following the core evaluation, participants may undergo selected scientific measurements for phenotyping purposes. Phenotyping measurements can occur over the course of several years.

Outcome Measures:

The study will use a wide variety of measurement tools for phenotyping purposes. These include: vital signs, medical history, physical exam, medical record review, qualitative pain interview, patient reported outcome measurements, psychological and behavioral measurements, clinical laboratory measurements, structural and functional imaging assessments using magnetic resonance imaging, and psychophysical measurements.

In summary, the NCCIH phenotyping protocol will enable investigators to obtain detailed clinical descriptions and collect phenotyping measurements from research participants, in particular those with pain disorders. It will collect information on research participants that, with consent, can be used to determine potential eligibility in other IRB-approved protocols and to support any further research and clinical decision making that would be based on this phenotyping information. The study will allow NCCIH investigators to perform descriptive research on pain disorders for use in hypothesis generation.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Are >= 12 years of age

EXCLUSION CRITERIA:

* Have difficulties with communication that make subjective pain assessment impossible or unreliable.
* Have acute medical or psychiatric health issues that create additional and substantial adverse risks related to study procedures. Medical examples are the acute complications of medical disease, such as asymptomatic hypertensive urgency, diabetic ketoacidosis, symptomatic hyperthyroidism, and unstable angina. Psychiatric examples are the acute complications of psychiatric disease, such as acute mania, paranoid delusions, or having acute panic attacks.
* Are participating in other ongoing research protocols such that phenotypic measurements would interfere with the conduct of an ongoing protocols or the receipt of a research treatment would influence the phenotypic measurements.
* Employees or staff that work at NCCIH.
* Pregnant women

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with or without pain disorders.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-07-22 (Actual); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-02-09 (Estimated)

PRIMARY OUTCOMES:
To enable for the deep, broad, and targeted phenotyping of individuals, in particular those with rare and unusual pain disorders. | 36 months
  Data are to be collected via medical history, physical examinations, questionnaires, laboratory samples and MRI imaging.

SECONDARY OUTCOMES:
To facilitate obtaining information relevant to determining potential eligibility in IRB-approved NIH protocols, in particular those of the Clinical Investigations Branch of NCCIH. | 36 months
  Data are to be collected via medical history, physical examinations, questionnaires, laboratory samples and MRI imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Backonja, M.D., Principal Investigator — National Center for Complementary and Integrative Health (NCCIH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We will only share deidentified data with repositories or publications, as specified in the protocol.

REFERENCES:
- [Derived] Amir C, Rose-McCandlish M, Weger R, Dildine TC, Mischkowski D, Necka EA, Lee IS, Wager TD, Pine DS, Atlas LY. Test-Retest Reliability of an Adaptive Thermal Pain Calibration Procedure in Healthy Volunteers. J Pain. 2022 Sep;23(9):1543-1555. doi: 10.1016/j.jpain.2022.01.011. Epub 2022 Feb 19. PMID 35189353
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-AT-0077.html